CLINICAL TRIAL: NCT01416545
Title: Children Education as Therapeutic Instrument for Cardiovascular Risk Reduction in Their Parents
Brief Title: Children Education and Cardiovascular Risk Reduction in Their Parents
Acronym: CETICARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Bruno Caramelli, Associated Professor of Cardiology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2009/17450-3
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Risk Reduction
Keywords: Primary Prevention; Cardiovascular disease; Child; Behavior modification; Activities, Educational
MeSH Terms: conditions — Risk Reduction Behavior; Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Active Comparator): Children received the same educational material for their parents and, additionaly, were exposed to a weekly educational program directed for cardiovascular prevention.
  Interventions: Behavioral: Educational program in cardiovascular prevention
- Control group (Placebo Comparator): The control group received written educational material directed for their parents and related to healthy lifestyle (nutrition, exercise and smoke quitting).
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Educational program in cardiovascular prevention — a weekly educational program in cardiovascular prevention with a multidisciplinary heath team during the year 2010. This intervention tried to teach to these children, in different manners appropriate for their age, concepts of healthy nutrition, avoidance of tobacco and physical activity. Both at the inclusion in the study and one year later we collect data of parents and their children of the two groups, in a single weekend, including nutritional and exercise survey, measures of weigh, height, waist circumference, arterial blood pressure, and laboratorial exams.
  Arms: Lifestyle counseling
Behavioral: Lifestyle counseling — The control group received written educational material directed for their parents and related to healthy lifestyle (nutrition, exercise and smoke quitting).
  Arms: Control group

SUMMARY:
This study aims to evaluate if a multidisciplinary educational program in primary cardiovascular prevention for children could improve the Framingham Score index of their parents after one year.

DETAILED DESCRIPTION:
Students aging 6 to 10 years old were exposed to two different approaches in the city of Sao Paulo, Brazil. For the students of the morning period (control group) we delivered written educational material for their parents in the beginning and middle of the year 2010 about healthy lifestyle (nutrition, exercise and smoke quitting). The students of the afternoon period (intervention group) received the same educational material for their parents and the children were exposed to a weekly educational program in cardiovascular prevention with a multidisciplinary heath team during the year 2010. This intervention tried to teach to these children, in different manners appropriate for their age, concepts of healthy nutrition, avoidance of tobacco and physical activity. Both at the inclusion in the study and one year later we collect data of parents and their children of the two groups, in a single weekend, including nutritional and exercise survey, measures of weigh, height, waist circumference, arterial blood pressure, and laboratorial exams.

ELIGIBILITY:
Inclusion Criteria:

* students aged 6 to 10 years old and their parents of a single private school of the city of Sap Paulo, Brazil

Exclusion Criteria:

* children and/or parents that do not agree to participate of the study;
* children and/or parents that are taking immunosupressive drugs;
* parents with known atherosclerotic disease such as angina or myocardial infaction, stroke, and/or peripheral arterial disease;
* parents with untreated hypothyroidism, untreated hypopituitarosm, nefrotic syndrome, chronic renal failure, congenital biliary allof, storage diseases, lupus and/oracquired immunodeficiency syndrome.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in cardiovascular risk measured by Framingham score index in parents whose children have participated (or not) in a multidisciplinary educational intervention for prevention of cardiovascular diseases. | Basal evaluation before intervention (basline) and one-year after intitiation of intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Caramelli, MD, PhD, Study Chair — University of Sao Paulo; Luciana S Fornari, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- InCor (Heart Institute) - Hospital das Clinicas da FMUSP, São Paulo, Brazil